CLINICAL TRIAL: NCT01180426
Title: The TOPAZ Study: A Long-Term Extension Study in Elderly Subjects With Relapsed/Refractory Acute Myeloid Leukemia to Allow Continued Therapy With Tosedostat
Brief Title: Extension Study With Tosedostat in Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chroma Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHR-2797-045
Record Dates: First submitted 2010-08-05; First posted 2010-08-12 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Relapse Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tosedostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tosedostat (Experimental)
  Interventions: Drug: CHR-2797

INTERVENTIONS:
Drug: CHR-2797 — 120mg once daily oral for 48 weeks

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy and safety profile of tosedostat in elderly patients suffering from refractory or relapsed Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
Extension protocol to the OPAL Study (CHR-2797-038).

Study mimics normal clinical practice; few procedures and visits are therefore mandated by the protocol. Timing of bone marrow assessment is also left at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent
* Completion of Visit 11 in the OPAL Study (Month 6 Visit)
* Investigator's opinion that the subject would benefit from continued therapy with tosedostat.

Exclusion Criteria:

* Any co-existing medical condition that in the Investigator's opinion will substantially increase the risk associated with the subject's participation in the study
* Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies
* Administration of any (other) investigational agent within 14 days of entry into TOPAZ.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of extended treatment with tosedostat | Protocol mandated visits every 12 weeks
  Primary outcome will be assessed using the following procedures/data:
  * Physical exams
  * Vital signs
  * Electrocardiography
  * Laboratory parameters (hematology, chemistry, urinalysis)
  * Adverse events
  * Serious adverse events

SECONDARY OUTCOMES:
Efficacy of extended treatment with tosedostat | Protocol-mandated visits every 12 weeks
  The secondary outcome will be assessed using the following parameters:
  * Overall survival
  * Relapse-free survival
  * Event-free survival
  * Clinical responses (Complete Remission, Complete Remission with Incomplete Platelet Recovery, Morphological Leukemia-Free State, Partial Remission, Stable Disease, Progressive Disease) including best response and time to response
  * Duration of clinical responses.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCLA Division of Hematology/Oncology, Los Angeles, California
  - University of Michigan, Ann Arbor, Michigan
  - John Theurer Cancer Center, Hackensack, New Jersey
  - New York Presbyterian Hospitacl, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson, Houston, Texas